CLINICAL TRIAL: NCT06569290
Title: Refinement and Testing of Recruitment Methodology for Behavioral Medication Adherence Interventions Using Behavioral Science-based Approaches
Acronym: STIC2IT-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Boston Medical Center (Other); Columbia University (Other)
Responsible Party: Principal Investigator, Niteesh K. Choudhry, MD, PhD, Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2024P002222; 5P30AG064199-05 (NIH)
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Diabetes; Pharmacist-Patient Relations; Medication Adherence
MeSH Terms: conditions — Diabetes Mellitus; Medication Adherence

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Principal investigators and data analysts will be masked to group assignment when analyzing data to determine the effectiveness of the recruitment strategy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Arm 1 (Active Comparator): Post card; control letter; 2 calls
  Interventions: Behavioral: Primer postcard; Behavioral: Control recruitment letter; Behavioral: 2 phone calls
- Arm 2 (Active Comparator): Post card; control letter; 4 calls
  Interventions: Behavioral: Primer postcard; Behavioral: Control recruitment letter; Behavioral: 4 phone calls
- Arm 3 (Active Comparator): Post card; behavioral letter; 2 calls
  Interventions: Behavioral: Primer postcard; Behavioral: Behavioral theory-informed recruitment letter (prospect theory); Behavioral: 2 phone calls
- Arm 4 (Active Comparator): Post card; behavioral letter; 4 calls
  Interventions: Behavioral: Primer postcard; Behavioral: Behavioral theory-informed recruitment letter (prospect theory); Behavioral: 4 phone calls
- Arm 5 (Active Comparator): No post card; control letter; 2 calls
  Interventions: Behavioral: Control recruitment letter; Behavioral: 2 phone calls
- Arm 6 (Active Comparator): No post card; control letter; 4 calls
  Interventions: Behavioral: Control recruitment letter; Behavioral: 4 phone calls
- Arm 7 (Active Comparator): No post card; behavioral letter; 2 calls
  Interventions: Behavioral: Behavioral theory-informed recruitment letter (prospect theory); Behavioral: 2 phone calls
- Arm 8 (Active Comparator): No post card; behavioral letter; 4 calls
  Interventions: Behavioral: Behavioral theory-informed recruitment letter (prospect theory); Behavioral: 4 phone calls

INTERVENTIONS:
Behavioral: Primer postcard — Inclusion of a mailed primer post card
  Arms: Arm 1; Arm 2; Arm 3; Arm 4
Behavioral: Control recruitment letter — a recruitment letter without any behaviorally-informed language
  Arms: Arm 1; Arm 2; Arm 5; Arm 6
Behavioral: Behavioral theory-informed recruitment letter (prospect theory) — the recruitment letter will use prospect theory and deliver a low risk, gain-framed behaviorally-informed message.
  Arms: Arm 3; Arm 4; Arm 7; Arm 8
Behavioral: 2 phone calls — 2 recruitment phone calls made by the call center
  Arms: Arm 1; Arm 3; Arm 5; Arm 7
Behavioral: 4 phone calls — 4 recruitment phone calls made by the call center
  Arms: Arm 2; Arm 4; Arm 6; Arm 8

SUMMARY:
The overarching goal of the proposed research is to prepare the clinical pharmacist intervention for sustainable implementation and dissemination. Because the effectiveness of the intervention has already been demonstrated in a NIH Stage Model IV trial, the investigators propose an Effectiveness-Implementation Type 3 Hybrid design, in which the primary focus is on testing different implementation methods, while secondarily observing clinical effects. The investigators' overarching hypothesis is to identify the most impactful elements of a behavioral theory-informed recruitment approach, which can be replicable across clinical settings.

Accordingly, the investigators propose to perform testing of a behaviorally-informed recruitment approaches in a community-based setting. Like the previous Tele-Pharmacy Intervention to Improve Treatment Adherence (STIC2IT) trial (NCT02512276), participants will be English or Spanish speaking adults ≥18 years of age identified through the electronic health record (EHR) as having poor disease control and/or poor medication adherence for diabetes. The primary care physicians of eligible patients identified through the EHR will be contacted to opt-out any patients they wish not to be included. Patients will then be randomized to each of the following conditions, such that there will be 8 total arms: (1) inclusion of a mailer primer (yes/no), (2) the most successful recruitment letter from the preliminary study using prospect theory (versus the control letter), and (3) intensity of the intervention outreach (4 calls vs. 2 calls). The investigators plan to enroll 584 participants who meet the inclusion criteria, with 73 patients per each of the 8 study arms.

Patients across all arms who agree to be scheduled will receive an appointment with one of the clinical pharmacists within the established BMC pharmacist program. The primary outcome will be completion of a clinical pharmacist appointment within 8 weeks after randomization. Key secondary outcomes will include scheduled visit rates, no-show rates for scheduled appointments, medication adherence over the 3-month follow-up, and clinical outcomes, including HbA1c levels measured using EHR data in the 3 months after randomization. The medication adherence and clinical outcomes will be used for the Aim 2 evaluation.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* English or Spanish speaking
* Receiving care from a BMC primary care provider
* Non-adherent to prescribed oral glucose-lowering medications as per pharmacy dispense records (proportion of days covered <80% to at least one eligible medication in last 6 months)
* Evidence of poor or worsening disease control

Exclusion Criteria:

* Evidence of terminal conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 584 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Completion of a clinical pharmacist adherence counseling appointment | within 8 weeks of receiving the intervention
  rate of participants who completed their clinical pharmacist consultation

SECONDARY OUTCOMES:
Schedule rates for clinical pharmacist adherence counseling appointment | within 8 weeks of receiving the intervention
  rate of participants who scheduled an appointment
No-show/cancellation rates | within 8 weeks of receiving the intervention
  rate of participants who did not show up to their appointment or cancelled their appointment after scheduling it
Glucose-lowering medication adherence | 3 months after randomization
  proportion of days covered of a glucose-lowering medication
Clinical outcome - HbA1c | 3 months after randomization
  HbA1c levels using EHR data

CONTACTS AND LOCATIONS:
Overall Officials: Niteesh K Choudhry, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No